CLINICAL TRIAL: NCT06792227
Title: Family-based Treatment at Home in Adolescents With Eating Disorders and Co-occurring Mental Health Conditions
Acronym: F-EET
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Responsible Party: Principal Investigator, Rik Knipschild, PhD, Karakter Kinder- en Jeugdpsychiatrie
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210-21
Record Dates: First submitted 2025-01-08; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders; Anorexia Nervosa; Eating Disorder Not Otherwise Specified
Keywords: Family Based Treatment; Youth; Eating Disorders; Anorexia Nervosa; Family Based Treatment at Home; FBT-H; FBT
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: To evaluate the effectiveness of FBT-H, we implemented a mixed-method approach combining a single-case design and a qualitative study. In the single-case design, 10 cases are intensively monitored throughout the FBT-H process, documenting interventions and their effects. The qualitative study complements this by gathering insights from adolescents, parents, and professionals about their experiences with FBT-H using structured interviews conducted separately with each group post-treatment to explore key topics. Together, these methods provide a comprehensive understanding of the impact of FBT-H.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mixed Methods Design (Experimental): To evaluate the effectiveness of FBT-H, we implemented a mixed-method approach combining a single-case design and a qualitative study. In the single-case design, 10 cases are intensively monitored throughout the FBT-H process, documenting interventions and their effects. The qualitative study complements this by gathering insights from adolescents, parents, and professionals about their experiences with FBT-H using structured interviews conducted separately with each group post-treatment to explore key topics. Together, these methods provide a comprehensive understanding of the impact of FBT-H.
  Interventions: Behavioral: FBT-H

INTERVENTIONS:
Behavioral: FBT-H — FBT is a structured treatment lasting 6-12 months, typically in an outpatient setting, with weekly sessions that gradually decrease in frequency over time (Lock & Le Grange, 2015). It empowers parents to manage their child's recovery from the ED. The first phase focuses on weight restoration, with parents responsible for all eating decisions and restricting physical activity to reduce ED's influence. In the second phase, eating responsibility gradually shifts back to the adolescent. The final phase supports healthy adolescent development as ED symptoms subside.
  The FBT-H adapts FBT to a home setting, with treatment led by family counselors and psychologists as part of a multidisciplinary team, including therapists, psychologists, a psychiatrist and a nurse specialist.

SUMMARY:
The significant impact of eating disorders on adolescents necessitates the evaluation of current treatments. Family-based Treatment (FBT) is the standard treatment but has modest remission rates, highlighting the need for improvements. Assessing its effectiveness in adolescents with co-occurring mental health conditions is also crucial. In the Netherlands, there is a growing focus on home-based treatment. This study aims to enhance remission rates in FBT by adapting it for use in a home setting (FBT-H).

DETAILED DESCRIPTION:
Background:

The significant impact of eating disorders on adolescents necessitates the evaluation of current treatments. Family-based Treatment (FBT) is the standard treatment but has modest remission rates, highlighting the need for improvements. Assessing its effectiveness in adolescents with co-occurring mental health conditions is also crucial. In the Netherlands, there is a growing focus on home-based treatment. This study aims to enhance remission rates in FBT by adapting it for use in a home setting (FBT-H).

Objective:

This mixed-method study combines single case studies with qualitative research. The primary objective is to assess the effects and experiences of FBT-H in adolescents with eating disorders and co-occurring mental health conditions across variables such as weight, eating disorder symptoms, anxiety, mood, well-being, quality of life, and family dynamics. Additionally, it explores the experiences of adolescents, parents, and practitioners with FBT-H.

Methods:

Adolescents (12-18 years old) with anorexia nervosa (AN) or other specified feeding or eating disorders (OSFED), alongside co-occurring mental health conditions, will participate in FBT-H, attending about two home sessions per week for 6-12 months. Ten patients will be monitored with intensive measurements over one year. Baseline assessments include somatic screening, clinical interviews, and evaluations of mood, anxiety, and family dynamics. The primary outcome is weight change from baseline to one year post treatment, and secondary outcomes (e.g., eating disorder symptoms, quality of life, parent-child relationships, and caregiving burden) are assessed at baseline and then every three months. General well-being and therapeutic relationships are tracked weekly. One-year post treatment, somatic health, and mood/anxiety symptoms will be reassessed alongside qualitative interviews with adolescents, parents, and practitioners.

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 12 to 18 years;
* meeting the criteria for AN or other specified feeding or eating disorder (OSFED);
* presence of co-occurring mental health conditions;
* sufficient command of the Dutch language by adolescents and parents;
* the family supports the treatment as a supportive system and is open to participating in the research.

Exclusion Criteria:

* acute suicidal behaviour requiring hospitalization within the 4 weeks prior to assessment for this study;
* cognitive limitations (IQ < 70);
* participation of a sibling in the current study (to prevent transfer of therapy effects between siblings);
* the adolescent does not receive tube feeding at the start of FBT-H and/or is not hospitalized due to an eating disorder at the start of treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Weight | Each session (week 1 - week 52, through study completion)
  Weight - each session The weight of the adolescent in kilograms (kg) is measured weekly to monitor progress. The weight is measured by an FBT-H practitioner in an FBT-H session. The weight is measured in the same way every week (e.g., in underwear). This is a standard measurement associated with the FBT intervention and takes approximately 5 minutes.

SECONDARY OUTCOMES:
Outcome Rating Scale | Each session (week 1 - week 52, through study completion)
  The ORS is a questionnaire in which participants indicate how they are doing in four components of their lives: personal, interpersonal, social, and general (Miller et al., 2003); translated by Hafkenscheid et al., 2003). These four components form the four items in this questionnaire, which can be answered on a scale from 0-10. There is a child and adult version of the ORS. A score of more to the left (0) indicates a negative score on the corresponding component, and a score of more to the right (10) indicates a more positive one. The internal consistency, measured by Cronbach's alpha, is .97 (26). Adolescents and their parents participating in this study will be asked to fill out this questionnaire at the beginning of each session, which requires approximately 1 minute.
Session Outcome Rating Scale | Each session (week 1 - week 52, through study completion)
  The SRS is a questionnaire in which adolescents express how they have experienced a session. The four items covered are relationship/contact, goals and topics, approach and method, and overall satisfaction. The SRS has the same setup as the previously mentioned ORS. The internal consistency, measured by Cronbach's alpha, is .88. Adolescents and parents participating in this study will be asked to fill out this questionnaire at the end of each treatment session, which takes approximately 1 minute.
Eating Disorder Examination Questionnaire | Adolescents in this study will complete the EDE-Q five times (T0 to T4)(T0 = Week 0, T1 = month 3, T2 = month 6, T3 = month 9, T4 = month 12) . It takes 10 minutes to complete the questionnaire.
  The EDE-Q is a self-report questionnaire used to assess the behaviours and characteristics of ED. The EDE-Q consists of a global scale (22 items) and four subscales: restraint, eating concern, weight concern, and shape concern. Each question can be answered on a scale from 1 to 6 or with a yes/no response. Satisfactory levels of internal consistency were observed.
Quality of Life | Adolescents and their parents are asked to complete this questionnaire five times (T0 to T4)(T0 = Week 0, T1 = month 3, T2 = month 6, T3 = month 9, T4 = month 12) and it requires 10 minutes to complete.
  Kidscreen-27 is a questionnaire measuring the quality of life of children in five dimensions: physical well-being, mental well-being, parent relations and autonomy, social support (from peers), and school situation. It consists of 27 questions, each of which has five answer options. Cronbach's alpha for all scales varies between average and good.
Parent-Child Interaction Questionnaire-Revised | The OKIV-R is administered a total of five times to both adolescents and their parents (T0 to T4)(T0 = Week 0, T1 = month 3, T2 = month 6, T3 = month 9, T4 = month 12) . The duration to complete the questionnaire is approximately10 minutes.
  The OKIV-R consists of questionnaires that measure how parents view the relationship with their child and how children view the relationship with their parents. The child-mother, child-father, and parent-child versions are available. It has 21 statements, and each statement has five answer options varying from never (1) to always (5). The revised version of the OKIV (OKIV-R) has high internal consistency.
Parenting Burden Questionnaire (Opvoedingsbelasting Vragenlijst (OBVL) | The OBVL is administered a total of five times to parents participating in this study (T0 to T4)(T0 = Week 0, T1 = month 3, T2 = month 6, T3 = month 9, T4 = month 12) , and it requires 15 minutes of their time.
  The OBVL is a questionnaire for parents about experiencing stress in parenting (Veerman et al., 2014).The OBVL consists of five scales (34 questions): parent-child relationship, parenting competence (7), depressive moods (7), role limitations (6), and health complaints (8). Each question has four answers that the parent can choose, varying from do not agree to totally agree. The scales of the OBVL have a reliability between .90 and .96 (McDonald's Omega).

CONTACTS AND LOCATIONS:
Locations (1):
- Karakter, Almelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to persmissions

REFERENCES:
- [Derived] Schapink AH, van der Velde J, Winkelhorst K, Kaijadoe S, Elgersma HJ, Le Grange D, Knipschild R, Klip H. Family-based treatment at home in adolescents with eating disorders and co-occurring mental health conditions: rationale and study design of a mixed methods trial. BMC Psychiatry. 2025 Apr 8;25(1):346. doi: 10.1186/s12888-025-06672-z. PMID 40200161